CLINICAL TRIAL: NCT04786054
Title: Genetic Association of Glucocorticoid Receptor Gene Polymorphisms With Binge Eating Disorders in Type 2 Diabetic Obese Female Adolescents
Brief Title: Genetic Association of Glucocorticoid Receptor Gene Polymorphisms With Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Dr Zainab Khan, Chief Resident, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: BEDCAI37628
Record Dates: First submitted 2021-02-26; First posted 2021-03-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Binge-Eating Disorder; Eating Disorders; Obesity; Diabetes Type 2; Adolescent Behavior
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders; Obesity; Diabetes Mellitus, Type 2; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BED (Active Comparator): Those who are diagnosed with having Binge Eating disorder. These individuals qualified after the questionnaire was administered.
  Interventions: Diagnostic Test: BED Questionnaire
- Group Non-BED (No Intervention): Those who are not diagnosed with having Binge Eating disorder

INTERVENTIONS:
Diagnostic Test: BED Questionnaire — BED Questionnaire
  Arms: Group BED

SUMMARY:
The aim of the present study was to specifically screen obese diabetic adolescent female individuals for BED, checking the variants of the GR gene (rs56149945; rs41423247) amongst identified individuals, and this led to assessing the impact of binge eating disorders on glycaemic control in obese diabetic adolescent females in Pakistan, South Asia.

DETAILED DESCRIPTION:
Challenges in eating for diabetic adolescents can be categorized as eating disorders (ED) and disordered eating symptoms (DES). Binge-eating disorder (BED) is defined as recurrent episodes of binge eating at least once a week over a three-month time period and it is accompanied by feeling the lack of control and marked distress over one's eating behaviour. The aim of the present study was to specifically screen obese diabetic adolescent female individuals for BED, checking the variants of the GR gene (rs56149945; rs41423247) amongst identified individuals, and this led to assessing the impact of binge eating disorders on glycaemic control in obese diabetic adolescent females in Pakistan, South Asia.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried females diagnosed with Type 2 diabetes > 12 months
* Age 10-19 years
* Obesity class I and II (based on BMI range of 30 - 40).

Exclusion Criteria:

* Presence of psychosis, major psychiatric or neurocognitive disorder
* Substance use
* Untreated attention-deficit hyperactivity disorder
* Use of psychopharmacological medications or psychotherapy
* Class III obesity

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Biological female
Enrollment: 91 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
BED | Baseline
  Presence of BED detected by individuals who score high on the BEDS7 Questionnaire administered

SECONDARY OUTCOMES:
NR3C1 Presence of variants of the GR gene (rs56149945; rs41423247) | Six months into the study after identifying all individuals who scored high on the BEDS7 Questionnaire
  Presence of variants of the GR gene (rs56149945; rs41423247)

CONTACTS AND LOCATIONS:
Locations (1):
- Zainab Khan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No